# BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU (FORM 3)

#### **LÜTFEN DİKKATLİCE OKUYUNUZ !!!**

Bu çalışmaya katılmak üzere davet edilmiş bulunmaktasınız. Bu çalışmada yer almayı kabul etmeden önce çalışmanın ne amaçla yapılmak istendiğini anlamanız ve kararınızı bu bilgilendirme sonrası özgürce vermeniz gerekmektedir. Size özel hazırlanmış bu bilgilendirmeyi lütfen dikkatlice okuyunuz, sorularınıza açık yanıtlar isteyiniz.

### ÇALIŞMANIN AMACI NEDİR?

Hijyenik ped ambalajı üzerindeki yazılı ve görsel mesajların kadınların aile planlamasına ilişkin bilgi ve tutumlarına etkisini belirlemek amacıyla planlanmıştır.

# KATILMA KOŞULLARI NEDİR?

Bu çalışmaya dahil edilme kriterleri;

- > 18-49 yaş aralığında,
- En az ilkokul mezunu olan,
- > 9-18 aylık bebeği olan,
- AP yöntemi kullanmayan veya geleneksel AP yöntemleri (geri çekme, takvim yöntemi),
- > Evli ve cinsel partneri mevcut olan,
- Aktif cinsel yaşamı olan,
- Düzenli menstrual siklusu olan,
- lletişimi engelleyen herhangi bir engeli olmayan,
- > Telefon numarasını vermeye gönüllü olan,
- > Akıllı telefon kullanan,
- > En az ilkokul mezunu olan kadınlar dahil edilecektir.

### NASIL BİR UYGULAMA YAPILACAKTIR?

Çalışma, müdahale grubu ve kontrol grubu olmak üzere iki gruptan oluşacaktır. Müdahale ve kontrol grubunda yer alan kadınlarla tanışılarak araştırmanın amacı ve çalışma planı hakkında bilgi verilecektir. Çalışmaya katılmayı kabul eden kadınların sözlü ve yazılı onamları alınacaktır. Daha sonra Kişisel Bilgi Formu'nun birinci bölümü yüz yüze görüşme tekniğiyle, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği kadının kendi bildirimine göre doldurulacaktır. İlk görüşme sonlandırılmadan önce kadına üç ay sonra telefon ile aranılacağı, online anket formun gönderileceği ve bunun doldurulması gerektiği bilgisi verilecektir. İkinci görüşmede, Tanıtıcı Bilgi Formu'nun ikinci bölümü, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği online anket form doldurma yöntemi aracılığıyla doldurulacaktır.

#### **SORUMLULUKLARIM NEDİR?**

Araştırma ile ilgili olarak sorulan sorulara tam ve yansız cevap vermeniz sizin sorumluluklarınızdır. Bu koşullara uymadığınız durumlarda araştırıcı sizi uygulama dışı bırakabilme yetkisine sahiptir.

### KATILIMCI SAYISI NEDİR?

| Girisimsel Olmayan Klinik Araştırmalar İçin Bilgilendirilmiş Gönüllü Olur | Belge Kodu | Rev. Tarihi / No.su: | Sayfa |
|---|---|---|---|
| Formu Strain Vitagen Hallar 15th Dilghertanning Schalla Star | Form 3 | 15.12.2016/ADÜSBF | 1/4 |

Araştırmaya, müdahale grubuna 50 kişi, kontrol grubuna 50 kişi olmak üzere toplam 100 kişi katılacaktır.

### **CALISMANIN SÜRESİ NE KADAR?**

Bu araştırma için öngörülen süre 12 aydır (Ekim 2022- Ekim 2023).

# GÖNÜLLÜNÜN BU ARAŞTIRMADAKİ TOPLAM KATILIM SÜRESİ NE KADAR?

Bu araştırmada yer almanız için öngörülen zamanınız 20-30 dakikadır.

### CALIŞMAYA KATILMA İLE BEKLENEN OLASI YARAR NEDİR?

Bu araştırma, hijyenik ped ambalajı üzerindeki yazılı ve görsel mesajların kadınların aile planlamasına ilişkin bilgi ve tutumlarına etkisini belirlemektir.

# ÇALIŞMAYA KATILMA İLE BEKLENEN OLASI RİSKLER NEDİR?

Beklenen risk yoktur.

# HERHANGİ BİR ZARARLANMA DURUMUNDA YÜKÜMLÜLÜK/SORUMLULUK KİMDEDİR VE NE YAPILACAKTIR?

Araştırmaya bağlı bir zarar söz konusu olduğunda, bu durumun tedavisi sorumlu araştırıcı tarafından yapılacak, ortaya çıkan masraflar araştırmacılar tarafından karşılanacaktır.

# ARAŞTIRMA SÜRESİNCE ÇIKABİLECEK SORUNLAR İÇİN KİMİ ARAMALIYIM?

Araştırma hakkında ek bilgiler almak için ya da çalışma ile ilgili herhangi bir sorun, istenmeyen etki ya da diğer rahatsızlıklarınız için 0534 259 50 88 no.lu telefondan Yasemin SÖKMEN'e başvurabilirsiniz.

# ÇALIŞMA KAPSAMINDAKİ GİDERLER KARŞILANACAK MIDIR?

Yapılacak araştırma masrafları size veya güvencesi altında bulunduğunuz resmi ya da özel hiçbir kurum veya kuruluşa ödetilmeyecektir.

#### ÇALIŞMAYI DESTEKLEYEN KURUM VAR MIDIR?

Çalışmanın etik kurul belgesi alındıktan sonra TÜBİTAK başvurusu yapılacaktır.

# ÇALIŞMAYA KATILMAM NEDENİYLE HERHANGİ BİR ÖDEME YAPILACAK MIDIR? Bu araştırmada yer almanız nedeniyle size hiçbir ödeme yapılmayacaktır.

# ARAŞTIRMAYA KATILMAYI KABUL ETMEMEM VEYA ARAŞTIRMADAN AYRILMAM DURUMUNDA NE YAPMAM GEREKİR?

Bu araştırmada yer almak tamamen sizin isteğinize bağlıdır. Araştırmada yer almayı reddedebilirsiniz ya da herhangi bir aşamada araştırmadan ayrılabilirsiniz; reddetme veya vazgeçme durumunda bile sonraki bakımınız garanti altına alınacaktır. Araştırmanın sonuçları bilimsel amaçla kullanılacaktır; çalışmadan çekilmeniz ya da araştırıcı tarafından çıkarılmanız durumunda, sizle ilgili tıbbi veriler bilimsel amaçla kullanılmayacaktır.

### KATILMAMA İLİŞKİN BİLGİLER KONUSUNDA GİZLİLİK SAĞLANABİLECEK MİDİR?

Size ait tüm tıbbi ve kimlik bilgileriniz gizli tutulacaktır ve araştırma yayınlansa bile kimlik bilgileriniz verilmeyecektir, ancak araştırmanın izleyicileri, yoklama yapanlar, etik kurullar ve resmi makamlar gerektiğinde tıbbi bilgilerinize ulaşabilir. Siz de istediğinizde kendinize ait tıbbi bilgilere ulaşabilirsiniz.

### Çalışmaya Katılma Onayı:

Yukarıda yer alan ve araştırmaya başlanmadan önce gönüllüye verilmesi gereken bilgileri gösteren 3 sayfalık metni okudum ve sözlü olarak dinledim. Aklıma gelen tüm soruları araştırıcıya sordum, yazılı ve sözlü olarak bana yapılan tüm açıklamaları ayrıntılarıyla anlamış bulunmaktayım.

| Girisimsel Olmayan Klinik Arastırmalar İçin Bilgilendirilmiş Gönüllü Olur | Belge Kodu | Rev. Tarihi / No.su: | Sayfa |
|---|---|---|---|
| Formu Singilia Singila | Form 3 | 15.12.2016/ADÜSBF | 2/4 |

Çalışmaya katılmayı isteyip istemediğime karar vermem için bana yeterli zaman tanındı. Bu koşullar altında, bana ait tıbbi bilgilerin gözden geçirilmesi, transfer edilmesi ve işlenmesi konusunda araştırma yürütücüsüne yetki veriyor ve söz konusu araştırmaya ilişkin bana yapılan katılım davetini hiçbir zorlama ve baskı olmaksızın büyük bir gönüllülük içerisinde kabul ediyorum. Bu formu imzalamakla yerel yasaların bana sağladığı hakları kaybetmeyeceğimi biliyorum.

Bu formun imzalı ve tarihli bir kopyası bana verildi.

| | GÖNÜLLÜNÜN | İMZASI |
|--------|------------|--------|
| ADI & | | |
| SOYADI | | |
| ADRESİ | | |
| TEL. & | | |
| FAKS | | |
| TARİH | | |

| VELAYET V | VEYA VESAYET ALTINDA BULUNANLAR İÇİN VELİ<br>VEYA VASİNİN | İMZASI |
|---|---|---|
| ADI & | | |
| SOYADI | | |
| ADRESİ | | |
| TEL. & | | |
| FAKS | | |
| TARİH | | |

| ARAŞT | TRMA EKİBİNDE YER ALAN VE YETKİN BİR<br>ARAŞTIRMACININ | İMZASI |
|--------|--------------------------------------------------------|--------|
| ADI & | | |
| SOYADI | | |
| TARİH | | |

| Girisimsel Olmayan Klinik Arastırmalar İçin Bilgilendirilmiş Gönüllü Olur | Belge Kodu | Rev. Tarihi / No.su: | Sayfa |
|---|---|---|---|
| Formu Singili Singil Si | Form 3 | 15.12.2016/ADÜSBF | 3/4 |

| | GEREKTİĞİ DURUMLARDA TANIK | İMZASI |
|--------|----------------------------|--------|
| ADI & | | |
| SOYADI | | |
| GÖREVİ | | |
| TARİH | | |

| Girişimsel Olmayan Klinik Araştırmalar İçin Bilgilendirilmiş Gönüllü Olur | Belge Kodu | Rev. Tarihi / No.su: | Sayfa |
|---|---|---|---|
| Formu | Form 3 | 15.12.2016/ADÜSBF | 4/4 |